CLINICAL TRIAL: NCT02337491
Title: Phase II Study of Pembrolizumab (MK-3475) With and Without Bevacizumab for Recurrent Glioblastoma
Brief Title: Pembrolizumab +/- Bevacizumab for Recurrent GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David Reardon, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-477
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Glioblastoma
Keywords: Recurrent
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: There is a safety lead-in before the start of the randomized phase 2 study.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A Safety Lead-In: Pembrolizumab (DL 0) + Bevacizumab (Experimental): Pembrolizumab (Dose Level 0): 200 mg administered intravenously on days 1 and 22 of each 42 day cycle Bevacizumab: 10 mg/kg administered Intravenously on days 1, 15 and 29 of each 42 day cycle
  Participants were treated until disease progression or unacceptable toxicity up to 16 cycles.
  Interventions: Drug: Pembrolizumab
- Cohort A: Pembrolizumab + Bevacizumab (Experimental): Pembrolizumab: 200 mg administered intravenously on days 1 and 22 of each 42 day cycle Bevacizumab: 10 mg/kg administered Intravenously on days 1, 15 and 29 of each 42 day cycle
  Participants were treated until disease progression or unacceptable toxicity up to 16 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab
- Cohort B: Pembrolizumab (Experimental): Pembrolizumab: 200 mg administered intravenously on days 1 and 22 of each 42 day cycle
  Participants were treated until disease progression or unacceptable toxicity up to 16 cycles.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: MK-3475; SCH 900475
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Cohort A: Pembrolizumab + Bevacizumab

SUMMARY:
In this research study, the investigators are looking to determine the effectiveness of Pembrolizumab (MK-3475) when given with bevacizumab or when given alone for the treatment of recurrent glioblastoma multiforme (GBM). This study will also test the safety and tolerability of Pembrolizumab (MK-3475) when given alone or with bevacizumab.

DETAILED DESCRIPTION:
Pembrolizumab (MK-3475) is a humanized monoclonal antibody. An antibody is a common type of protein made in the body in response to a foreign substance. Antibodies attack foreign substances and protect against infection. Antibodies can also be produced in the laboratory for use in treating patients, an antibody that is made in the lab is also known as a humanized monoclonal antibody. There are now several approved antibodies for the therapy of cancer and other disease. Pembrolizumab (MK-3475) has been studied in lab experiments and in other types of cancer. Information from these studies suggests that Pembrolizumab (MK-3475) may be beneficial in your type of cancer. Bevacizumab, also known as Avastin, is approved by the FDA for treating recurrent GBM. Bevacizumab is an anti-angiogenic medicine, which means it blocks blood vessels from forming that could supply the tumor with nutrients and oxygen.

There is a safety lead-in to evaluate pembrolizumab in combination of with bevacizumab (cohort A) expected to enroll up to 18 participants. Three dose levels (DL) are evaluated for pembrolizumab administered at 200 mg (flat dosing) under various dose intervals: every 3 (DL 0), 4 (DL -1) or 6 (DL -2) weeks. A standard 3+3 design is used starting at DL 0. De-escalation may occur depending on observation of dose-limiting toxicity (DLT). At least 6 participants will be evaluated for DLT at DL 0. The Phase II study randomizes participants to cohort A: pembrolizumab (using the MTD determined in the safety lead-in) and bevacizumab or cohort B: pembrolizumab monotherapy (using the MTD determined in the safety lead-in). Accrual goals are established for each cohort: A n=50 and B n=30 participants. The two cohorts are evaluated independently against a historical control and not compared. All participants treated at the safety lead-in established MTD dose level will be rolled into the Phase II cohort.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma). Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made.
* Previous first line therapy with at least radiotherapy and temozolomide
* Be at first or second relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* CT or MRI within 14 days prior to start of study drug.
* An interval of at least 4 weeks (to start of study agent) between prior surgical resection or one week for stereotactic biopsy.
* An interval of at least 12 weeks from the completion of radiation therapy to start of study drug unless there is a new area of enhancement consistent with recurrent tumor outside the radiation field or there is unequivocal histologic confirmation of tumor progression
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* From the projected start of scheduled study treatment, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency.
* Has tumor primarily localized to the brainstem or spinal cord.
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Has received systemic immunosuppressive treatments within 6 months of start of study drug
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 4 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of start of study drug.
* Has received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or convection enhanced delivery.
* Requires therapeutic anticoagulation with warfarin at baseline; patients must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to starting study drug; however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed.
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug
* Has evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans.
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of start of study drug.
* Has a known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial
* Has a known history of HIV
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Has a known hypersensitivity to any of the study therapy products.
* Has received anti-angiogenic or anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc)
* Has a history of non-healing wounds or ulcers, or bone refractures within 3 months of fracture
* Has a history of arterial thromboembolism within 12 months of start of study drug.
* Has inadequately controlled hypertension
* Has a history of hypertensive crisis or hypertensive encephalopathy
* Has had clinically significant cardiovascular disease within 12 months of start of study drug
* Has a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UT, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] de Melo SM, Elias Nunes da Silva ME, Torloni MR, Riera R, De Cicco K, Latorraca CO, Pinto ACPN. Anti-PD-1 and anti-PD-L1 antibodies for glioma. Cochrane Database Syst Rev. 2025 Jan 8;1(1):CD012532. doi: 10.1002/14651858.CD012532.pub2. PMID 39777725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between Feb 2015 and June 2016
Period: Overall Study
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
Started | 50 | 30
Completed | 0 | 0
Not Completed | 50 | 30
Not completed — Death | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Progressive Disease | 44 | 28
Not completed — On Treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab | Total
Number analyzed (Participants) | 50 | 30 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.7) | 51.8 (13.3) | 51.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 35 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 41 | 24 | 65
  Unknown or Not Reported | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pembrolizumab Maximum Tolerated Dose (MTD) [Cohort A Safety Lead-In]
Description: The MTD of pembrolizumab in combination with bevacizumab 10 mg/kg intravenously (IV) on days 1, 15 and 29 of each 42 day cycle is determined by the number of participants who experience a dose limiting toxicity (DLT) at the various regimens of dosing frequency of pembrolizumab 200 mg IV administered under evaluation. See subsequent primary outcome measure for the DLT definition. The MTD is defined as the pembrolizumab dose frequency regimen at which fewer than one-third of participants experience a DLT. If de-escalation does not occur per design, then the starting dose is the Recommended Phase II Dose (RP2D).
Time Frame: one cycle/42 days
Population: The analysis dataset is comprised of all participants who enrolled in the safety lead-in study. Only dose level 0 was evaluated and no de-escalation doses were evaluated.
Measure: Number; unit: mg every 3 weeks
Arm/Group | Cohort A Safety Lead-In: Pembrolizumab (DL 0) + Bevacizumab
Number analyzed (Participants) | 6
mg every 3 weeks | 200

2. Primary Outcome: Pembrolizumab Dose Limiting Toxicity (DLT) [Cohort A Safety Lead-In]
Description: A DLT is defined as an adverse event (AE) that (a) is >= grade 3 and related to the pembrolizumab with an attribution of possible, probably or definite, and (b) occurs during and/or begins during the first 42 days of study treatment, and (c) does not meet any of the following exception criteria: grade 3 immune-related AE that downgrades to <= grade 2 within 5 days, or <= grade 1/baseline within 14 days of onset; grade 3 asymptomatic endocrinopathy; grade 3 inflammatory reaction attribution to anti-tumor response; grade 3 pneumonitis, neurologic event, or uveitis that downgrades to <=grade 1 within 3 days; liver transaminase elevation <= 8 times institutional upper limit of normal (ULN); total bilirubin <= 5 times institutional ULN; any pre-existing lab abnormality that deteriorates to grade 3/4 and determine not clinically significant by Investigator, Overall Principal Investigator and Sponsor.
Time Frame: The evaluation for MTD occurred continuously through one cycle of treatment (42 days).
Population: The analysis dataset is comprised of all participants who enrolled in the safety lead-in study.
Measure: Number; unit: participants with DLT
Arm/Group | Cohort A Safety Lead-In: Pembrolizumab (DL 0) + Bevacizumab
Number analyzed (Participants) | 6
participants with DLT | 0

3. Primary Outcome: 6-Month Progression-Free Survival (PFS6)
Description: PFS6 is the proportion of patients remaining alive and progression-free at 6-months from study entry.
  Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria. PD is a >25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition.
Time Frame: Disease was assessed radiographically for response every cycle on treatment. Treatment duration in cycles (cycle=42 days) was a mean (SD) of 4.5 (4.4) for Cohort A and 2.5 (2.7) for Cohort B. Assessment at week 72/cycle 12 pertains to the 6-month PFS.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 50 | 30
proportion of participants | 0.26 [0.146 to 0.403] | 0.067 [0.009 to 0.221]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on Kaplan-Meier is defined as the time from study entry to the earliest documentation of disease progression (PD) or death. Participants alive without evidence of PD were censored at the date of last disease assessment. Per Response Assessment in Neuro-Oncology (RANO) criteria, PD is a >25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition.
Time Frame: Disease was assessed radiographically for response every cycle on treatment and every 6 weeks long-term. Median PFS follow-up (months) was 25 for Cohort A and 26 for Cohort B.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 50 | 30
months | 4.1 [2.8 to 5.5] | 1.4 [1.4 to 2.7]

5. Secondary Outcome: Overall Survival (OS)
Description: OS based on Kaplan-Meier is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival every 3 months from the end of treatment until death or lost to follow-up. Median survival follow-up was 25 months for each cohort.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 50 | 30
months | 8.8 [7.7 to 14.2] | 10.3 [8.5 to 12.5]

6. Secondary Outcome: Overall Radiographic Response (ORR)
Description: ORR was established based on Response Assessment in Neuro-Oncology (RANO) criteria. RANO criteria has 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown. CR: disappearance of all enhancing lesions, stable or improved non-enhancing lesions, and stable or improved clinically. PR: >= 50% decrease in sum of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, stable or improved non-enhancing lesions, and stable or improved clinically. PD: >25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition. SD: does not qualify for CR, PR or PD.
Time Frame: Disease was assessed radiographically for response every cycle on treatment. Treatment duration in cycles (each cycle=42 days) was a mean (SD) of 4.5 (4.4) for Cohort A and 2.5 (2.7) for Cohort B.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 50 | 30
percentage of participants | 0.20 [0.11 to 0.32] | 0.0 [0.0 to 0.095]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment for unresolved AEs and up to day 90 for serious adverse events. AEs were evaluated over treatment which was a maximum duration of 16 cycles (approximates 22 months).
Description: SAEs defined per protocol and all remaining AEs categorized as Other AE without regard to treatment attribution.
Groups:
- Cohort B: Pembrolizumab: Pembrolizumab (Dose Level 0): 200 mg administered intravenously on days 1 and 22 of each 42 day cycle
  Participants were treated until disease progression or unacceptable toxicity up to 16 cycles.
Arm/Group | Cohort A: Pembrolizumab + Bevacizumab | Cohort B: Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/50 | 1/30
Serious Adverse Events (participants affected / at risk) | 22/50 | 10/30
Other Adverse Events (participants affected / at risk) | 50/50 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Pembrolizumab + Bevacizumab (N=50) | Cohort B: Pembrolizumab (N=30)
Alanine aminotransferase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 1
Edema cerebral (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 3 | 1
Lethargy (Nervous system disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 6 | 2
Thromboembolic event (Vascular disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular disorders - Other (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Pembrolizumab + Bevacizumab (N=50) | Cohort B: Pembrolizumab (N=30)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Agitation (Psychiatric disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 8 | 2
Alkaline phosphatase increased (Investigations) | 3 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 5 | 4
Anorgasmia (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 2
Aspartate aminotransferase increased (Investigations) | 9 | 0
Ataxia (Nervous system disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 1
Blurred vision (Eye disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0
Cardiac troponin T increased (Investigations) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 2 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 5 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 2 | 0
Confusion (Psychiatric disorders) | 9 | 7
Conjunctivitis (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Creatinine increased (Investigations) | 4 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 12 | 1
Dizziness (Nervous system disorders) | 7 | 1
Dry eye (Eye disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 1
Dysphasia (Nervous system disorders) | 11 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema face (General disorders) | 2 | 0
Edema limbs (General disorders) | 3 | 5
Endocrine disorders - Other (Endocrine disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 6 | 3
Eye infection (Infections and infestations) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Facial muscle weakness (Nervous system disorders) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 5
Fatigue (General disorders) | 21 | 12
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 3 | 1
Flu like symptoms (General disorders) | 2 | 1
Flushing (Vascular disorders) | 1 | 0
Gait disturbance (General disorders) | 10 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 2
Headache (Nervous system disorders) | 21 | 16
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 28 | 2
Hyperthyroidism (Endocrine disorders) | 5 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 10 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 5 | 2
Immune system disorders - Other (Immune system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 2
Investigations - Other (Investigations) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 7 | 3
Malaise (General disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 6 | 4
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 15 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 7 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 6
Neuralgia (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 10 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Oral hemorrhage (Gastrointestinal disorders) | 3 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Palpitations (Cardiac disorders) | 3 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Paresthesia (Nervous system disorders) | 6 | 3
Penile infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 10 | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Proteinuria (Renal and urinary disorders) | 9 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Psychiatric disorders - Other (Psychiatric disorders) | 2 | 1
Psychosis (Psychiatric disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Rash pustular (Infections and infestations) | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Seizure (Nervous system disorders) | 11 | 4
Sinus bradycardia (Cardiac disorders) | 3 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 13 | 0
Skin infection (Infections and infestations) | 4 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 6 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0
Vascular disorders - Other (Vascular disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 3
Weight loss (Investigations) | 5 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 12 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No